CLINICAL TRIAL: NCT04044443
Title: Post Market Registry of the IMPEDE and IMPEDE-FX Embolization Plugs
Brief Title: IMPEDE and IMPEDE-FX Embolization Plug Registry
Acronym: EMBO-PMS
Status: Active, not recruiting | Type: Observational
Sponsor: Shape Memory Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD1012
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Vascular Embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: IMPEDE, IMPEDE-FX or IMPEDE-FX RapidFill — Peripheral vascular embolization

SUMMARY:
EMBO-PMS is a prospective, multicentre, registry study of the IMPEDE and IMPEDE-FX Embolization Plug Systems

ELIGIBILITY:
Inclusion Criteria:

* Study participant is ≥18 years of age
* Study participant is considered a candidate for arterial or venous embolization of the peripheral vasculature

Exclusion Criteria:

* Study participant has an inability to provide written informed consent
* Study participant/treatment outside of the approved study device labeling, instructions for use (IFU)
* Study participant is a prisoner or member of other vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult study participants considered candidates for a peripheral vascular embolization procedure
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety - Rate of freedom from serious adverse events | 30 days
  Rate of freedom from serious adverse events related to the study devices and/or procedure, per review and adjudication by medical monitor
Efficacy - Rate of technical success (embolization of target vessel) | Immediately after the intervention
  Technical success, defined as embolization of the target area after deployment of the study device

SECONDARY OUTCOMES:
Efficacy - Rate of recurrence of clinical symptoms, based on original complaint | 90 days
  Number of participants free of recurrent clinical symptoms, based on clinical symptoms of original complaint
Efficacy - Rate of treated vessel occlusion | 90 days
  Treated vessel occlusion, measured per study site standard of care for the original condition treated
Safety - Rate of freedom from serious adverse events | 90 days
  Rate of freedom from serious adverse events related to the study devices and/or procedure, per review and adjudication by medical monitor

CONTACTS AND LOCATIONS:
Overall Officials: Robert Morgan, MBChB, Study Chair — St George's Hospital (St George's University Hospitals NHS Foundation Trust); Götz Richter, Study Chair — Klinikum Stuttgart
Locations (10):
- Germany (8):
  - Universitätsklinikum Carl-Gustav-Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein (Campus Kiel), Kiel
  - UNIVERSITÄTSKLINIKUM LEIPZIG AöR, Leipzig
  - Klinikum München rechts der Isar, München
  - Klinikum Nürnberg, Nuremberg
  - Klinikum StuttGart, Stuttgart
  - Uniklinikum Würzburg, Würzburg
- United Kingdom (2):
  - St George's Hospital (St George's University Hospitals NHS Foundation Trust), London
  - St Mary's Hospital (Imperial College Healthcare NHS Trust), London

IPD SHARING:
Plan to Share IPD: No